CLINICAL TRIAL: NCT06983730
Title: Development of a Clinical Experimental Heat Stress Protocol and Exploration of the Effect of Niacinamide on Physiologic, Metabolic, and Biochemical Responses to Heat Stress
Brief Title: The Kidney's Response to Exercise in Heat, and the Impact of Vitamin B3 on This Response
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Boston University Charles River Campus (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Nathan Raines, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2024P000637; K23DK138320 (NIH)
Record Dates: First submitted 2025-05-14; First posted 2025-05-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Heat Strain; Healthy Volunteer Study; Kidney Dysfunction
Keywords: NAD+; Niacinamide; Vitamin B3; Experimental heat strain
MeSH Terms: interventions — Niacinamide

STUDY DESIGN:
Intervention Model Description: There are two phases to this study. The first phase is a dose-response phase evaluating the effect of experimental heat strain on kidney metabolic and stress response. The second phase uses this experimental heat strain at a dose producing kidney metabolic and stress response to conduct a crossover trial investigating how Vitamin B3 impacts the kidney's metabolic and stress response during heat strain.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin B3, then placebo (Experimental): Individuals will receive 1000mg oral Vitamin B3 daily for two days leading up to their first exercise session, and oral placebo daily for two days leading up to their second exercise session.
  Interventions: Dietary Supplement: Vitamin B3
- Placebo, then vitamin B3 (Experimental): Individuals will receive 1000mg oral placebo daily for two days leading up to their first exercise session, and oral vitamin B3 daily for two days leading up to their second exercise session.
  Interventions: Dietary Supplement: Vitamin B3

INTERVENTIONS:
Dietary Supplement: Vitamin B3 — 1000mg once a day orally for two days, once the day before the exercise session, and once the day of the exercise session.
  Other Names: niacinamide

SUMMARY:
The goal of this clinical trial is to learn about the processes occurring in the kidneys while under heat stress in healthy volunteers. The main questions it aims to answer are:

* How do the chemicals produced by the body change under conditions of higher versus lower heat stress?
* What role does a specific area of the body's metabolism, known as NAD+ metabolism, play in the body's response to heat stress, and can this response be modified by taking vitamin B3?

DETAILED DESCRIPTION:
To answer these questions, researchers will compare the chemical changes in each participant under progressively higher levels of heat stress, and while taking either vitamin B3 or a placebo.

This clinical trial will occur in two stages. Participants may choose participate in stage 1 only, stage 2 only, or both parts of this clinical trial.

During stage 1, participants will exercise using a stationary rowing ergometer in a hot and humid environmental chamber for three sessions, each session separated by about a week.

* Each session, they will be asked to work out at a progressively higher intensity with climate conditions kept the same in the chamber.
* More intense exercise produces greater heat stress, resulting in lower, moderate, and higher levels of heat stress exposure across the three sessions.
* Researchers will see how chemicals in the blood and urine, along with physical measurements like heart rate and body temperature, change across these different levels of heat stress.

During stage 2, participants will exercise using the same rowing ergometer in the same environmental chamber. They will do this for two sessions, each separated by about a week.

* One of the sessions each participant will take vitamin B3, and the other session each participant will take placebo.
* Heat stress exposure will be the same each session.
* Researchers will again see how chemicals in the blood and urine, along with physical measurements like heart rate and body temperature, differ between sessions with vitamin B3 and sessions with placebo

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Any race
* Estimated glomerular filtration rate greater than 90 ml/min/1.73m2
* Urine albumin/creatinine ratio less than 30mg/g
* Nonsmoker
* No regular dietary supplements, particularly vitamin B3
* Physically fit, defined as having a VO2 max of between 35 and 60mL/kg/min

Exclusion Criteria:

* Medical condition preventing safe participation in exercise during heat
* Allergy to Vitamin B3
* Severe food allergies or dietary restrictions that would preclude eating the planned study diet without major modifications

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Urinary neutrophil gelatinase-associated lipocalin | Pre- and immediately post- heat stress exposure
  Marker of stress and injury in the kidney
Urinary TIMP2 (tissue inhibitor of metalloproteinase-2) and IGFBP7 (insulin-like growth factor-binding protein 7) | Pre- and immediately post- heat stress exposure
  Marker of kidney stress and injury

SECONDARY OUTCOMES:
Urine Quinolinate to Tryptophan Ratio | Pre- and immediately post- heat stress exposure
  Ratio of quinolinate to tryptophan in the urine
Serum creatinine | Pre- and immediately post- heat stress exposure
  Marker of kidney function

OTHER OUTCOMES:
Urine and serum metabolites, including metabolites related to nicotinamide adenine dinucleotide (NAD+) | Pre-, during, immediately post, and 24 hours post- heat stress exposure
  Other chemical byproducts of metabolism and exposure that may change during or impact the effect of heat stress, measured using mass spectrometry
Urine and serum nicotinamide levels | Pre-, during, immediately post, and 24 hours post- heat stress exposure
  Levels of the interventional supplement, vitamin B3 (nicotinamide)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan H Raines, MD MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Boston University, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be stored in the Harvard Dataverse Repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data availability will begin at the time of an associated publication or the end of the performance period, whichever comes first. Data will continue to be available for ten years after completion of study activities.
Access Criteria: Researchers may request controlled-access data using standard processes at the repository.
URL: https://dataverse.harvard.edu/